CLINICAL TRIAL: NCT02379494
Title: First Trimester Prediction of Preeclampsia and Fetal Growth Restriction Using Uterine Artery Doppler, Maternal Blood Pressure, Maternal Characteristics, Placental Volume and Maternal Serum Factors
Brief Title: First Trimester Prediction of Preeclampsia and Fetal Growth Restriction
Status: Completed | Type: Observational
Sponsor: Fetal Medicine Foundation (Other)
Collaborators: Wright State University (Other)
Responsible Party: Sponsor
Other Study IDs: SC#5031
Record Dates: First submitted 2014-02-20; First posted 2015-03-05 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2016-02

CONDITIONS: Preeclampsia; Fetal Growth Restriction
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A 5cc maternal blood sample will be obtained through standard blood draw. The blood will first be transferred onto a dry blood requisition form card. The blood sample will be refrigerated and the serum and dried blood spot samples will be sent to Perkin Elmer Laboratories (see attachment C for collection protocols). The maternal serum levels of PAPP-A, PLGF, AFP, and free β hCG will be measured according to a protocol established by Perkin Elmer Laboratories.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate the feasibility of screening for preeclampsia and fetal growth restriction between 11-13+6 weeks' gestation utilizing the combination of uterine artery doppler, maternal blood pressure, maternal characteristics, placental volume, and maternal serum factors, including PAPPA-A, PLGF, AFP and free Beta HCG. This is a non interventional study.

DETAILED DESCRIPTION:
Preeclampsia (PE) is a condition which affects approximately 2% of all pregnancies and can be a major cause of maternal and perinatal morbidity/mortality (2). The suspected underlying mechanism of PE is thought to be impaired trophoblastic invasion of the maternal spiral arteries leading to impaired placental perfusion, placental ischemia and subsequent development of endothelial dysfunction (3). There is evidence that PE, which is commonly associated with fetal growth restriction, can be predicted effectively at 11-13 weeks gestational age by combined screening algorithms combining uterine artery pulsatility index (PI), maternal mean arterial pressure (MAP) and maternal serum concentrations of placental products including but not limited to plasma protein A (PAPP-A), and placental growth factor (PLGF) (4-6).

Aim of Study/Hypothesis:

The aim of this study is to develop an algorithm based on the combination of maternal factors, uterine artery pulsatility index, mean arterial pressure, placental volume and serum biomarkers to estimate patient specific risks for the development of Preeclampsia in a US population.

ELIGIBILITY:
Inclusion Criteria:

All patients during their first trimester visit

Exclusion Criteria:

Fetal anomalies Pregnancies ending in termination, miscarriage or fetal death prior to 22 weeks and cases with no pregnancy follow up.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All pregnant patients during their first trimester
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2013-03; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Development of Preeclampsia | During the first trimester (11-13+6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jiri D Sonek, MD, Principal Investigator — Fetal Medicine Foundation/USA
Locations (1):
- Miami Valley Hospital, Dayton, Ohio, United States